CLINICAL TRIAL: NCT00079664
Title: Tai Chi Training and Sleep Enhancement in the Elderly
Brief Title: Comparing Tai Chi Training to a Low-Stress Physical Activity to Enhance Sleep in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03MH062327 (NIH); R03MH062327 (NIH); DSIR AT-SO
Record Dates: First submitted 2004-03-10; First posted 2004-03-12 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Sleep Deprivation; Sleep Initiation and Maintenance Disorders
Keywords: Tai Ji
MeSH Terms: conditions — Sleep Deprivation; Sleep Initiation and Maintenance Disorders | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Tai Chi

SUMMARY:
The purpose of this study is to examine the effects of Tai Chi, in comparison to conventional exercise, on the quality of sleep among sedentary older adults.

DETAILED DESCRIPTION:
Elderly individuals often suffer from sleep disturbances. Chronic sleep problems can cause significant medical, psychological, and social disruptions. Although many sleep-related studies exist, few studies have focused on improving quality of sleep. Tai Chi, an exercise that incorporates meditation and breathing with whole body movements, may improve the quality of sleep and health status of elderly individuals.

Participants will be randomly assigned to either a Tai Chi group or a conventional exercise control group. Participants in each group will exercise for 60 minutes, 3 times per week, for 6 months. Assessment of sleep quality and health status will be done at study start, 3 months, 6 months, at the end of the study, and at a 3-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary, as defined by a lack of regular exercise during the previous 6 months
* Healthy to the degree that participation in exercise testing and an exercise program would not exacerbate any existing disease condition
* Physician's clearance for participation
* Willingness to adhere to the conditions of the study

Exclusion Criteria:

* Sleep medication or other psychotropic medication during the study
* Current sleep disorder treatment
* Significant cognitive impairment as indicated by a score of 3 on the Pfeiffer Mental Status Questionnaire
* More than 7 alcoholic beverages per week or use of alcohol close to bedtime
* Smoking more than 10 cigarettes per day
* Score of 5 or higher in the Pittsburgh Sleep Quality Index questionnaire
* Score of 3 or higher on 2 out of 3 sleep items drawn from the Sleep Questionnaire and Assessment of Wakefulness

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-09; Primary Completion 2002-03 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States